CLINICAL TRIAL: NCT00842959
Title: Check of Optical Features and Accuracy of the Zeiss ZO Lens of the Company Carl Zeiss Meditec After Selection and Calculation With OKULIX
Brief Title: Check of Optical Features and Accuracy of the Zeiss ZO Lens After Selection and Calculation With OKULIX
Acronym: ZO Okulix
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Andreas Langer, Acri.Tec GmbH
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: Acri.Tec-RES-DE-273
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Cataract
Keywords: Improvement of adjustment accuracy of intraocular lenses and imaging quality
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZO (Other): XL Stabi ZO or Invent ZO
  Interventions: Device: Invent ZO; Device: XL Stabi ZO

INTERVENTIONS:
Device: Invent ZO — monofocal aspheric IOL for implantation into capsular bag
Device: XL Stabi ZO — monofocal aspheric IOL for implantation into capsular bag

SUMMARY:
It is planned to implant the intraocular lenses XL Stabi ZO and Invent ZO into the eyes of patients for whom a cataract operation is medically indicated. The lenses are marketed and CE certified. Their implantation is clinical routine.

In the trial the accuracy of prediction of target refraction and the difference between calculated and measured contrast vision will be examined for both lens types.

ELIGIBILITY:
Inclusion Criteria:

* Indication for cataract operation
* Written informed consent of patient after information

Exclusion Criteria:

* Immobility
* Limited capacity of understanding
* Diseases that hamper a follow-up examination
* Astigmatism >2.0 D
* Patients with ocular diseases who may be expected to show a vision of less than 0.63 (decimal) two months after cataract surgery with implantation of intraocular lens
* Complications during surgery, especially complications with positioning of the intraocular lens and with capsulorhexis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of prediction of target refraction | postop.
Difference between calculated and measured contrast vision. | postop.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Wahl, MD, Principal Investigator — Universitäts-Augenklinik Mainz
Locations (1):
- Universitäts-Augenklinik Mainz, Mainz, Germany